CLINICAL TRIAL: NCT01556438
Title: A Phase 1 Study of Tabalumab (LY2127399) in Combination With Bortezomib and Dexamethasone in Japanese Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Study of Tabalumab (LY2127399) in Japanese Participants With Relapsed or Refactory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14459; H9S-JE-JDCI (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-03-15; First posted 2012-03-16 (Estimated); Results first posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2018-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — tabalumab; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 100 mg Tabalumab+Bortezomib (BTZ)IV+Dexamethasone (Dex) (Experimental): Cohort 1. 100 mg tabalumab (LY2127399) intravenously (IV) on day 1 of each cycle, each cyle is 21 days. Bortezomib (BTZ), 1.3 milligram per square meter (mg/m^2), IV on days 1, 4, 8, 11 of Cycle 1-8, then on days 1, 8, 15, 22 from Cycle 9 onward. Oral dexamethasone (Dex), 20 mg/day, on day of and day after BTZ.
  Interventions: Biological: Tabalumab; Drug: Bortezomib IV; Drug: Dexamethasone
- 300 mg Tabalumab+BTZ IV+Dex (Experimental): Cohort 2. 300 mg tabalumab (LY2127399) IV on day 1 of each cycle, each cycle is 21 days. BTZ, 1.3 mg/m^2, IV on days 1, 4, 8, 11 of Cycle 1-8, then on days 1, 8, 15, 22 from Cycle 9 onward. Oral dex, 20 mg/day, on day of and day after BTZ.
  Interventions: Biological: Tabalumab; Drug: Bortezomib IV; Drug: Dexamethasone
- 300 mg Tabalumab+BTZ SC+Dex (Experimental): Cohort 2-SC. 300 mg tabalumab (LY2127399)IV on day 1 of each cycle, each cycle is 21 days. BTZ, 1.3 mg/m^2, subcutaneously (SC) on days 1, 4, 8, 11 of Cycle 1-8, then on days 1, 8, 15, 22 from Cycle 9 onward. Oral dex, 20 mg/day, on day of and day after BTZ. Cohort 2-SC was added per protocol amendment in February 2013.
  Interventions: Biological: Tabalumab; Drug: Bortezomib SC; Drug: Dexamethasone

INTERVENTIONS:
Biological: Tabalumab — Administered IV
  Other Names: LY2127399
Drug: Bortezomib IV — Administered IV
  Arms: 100 mg Tabalumab+Bortezomib (BTZ)IV+Dexamethasone (Dex); 300 mg Tabalumab+BTZ IV+Dex
Drug: Bortezomib SC — Administered SC
  Arms: 300 mg Tabalumab+BTZ SC+Dex
Drug: Dexamethasone — Administered orally

SUMMARY:
The purpose of this study is to evaluate the safety and effect on the body of Tabalumab (LY2127399) in combination with bortezomib and dexamethasone in Japanese participants with relapsed or refractory multiple myeloma (MM).

DETAILED DESCRIPTION:
The study has 3 cohorts. Cohort 2 and cohort 2-SC will be conducted in parallel with some data presented combined.

Cohort 1 - Participants will receive 100 mg Tabalumab (LY2127399) intravenously (IV), 1.3 milligram per square meter (mg/m^2) bortezomib IV, and 20 mg dexamethasone orally.

Cohort 2 - Participants will receive 300 mg Tabalumab (LY2127399) IV, 1.3 mg/m^2 bortezomib IV, and 20 mg dexamethasone orally.

Cohort 2-SC - Participants will receive 300 mg Tabalumab (LY2127399) IV, 1.3 mg/m^2 bortezomib subcutaneously (SC), and 20 mg dexamethasone orally.

Cohort 2-SC was added per protocol amendment in February 2013.

ELIGIBILITY:
Inclusion Criteria:

* Have relapsed or refractory MM treated with at least 1 prior regimen. Prior therapy with bortezomib is allowed if there was previously at least a minimal response (MR).
* Have measurable disease as defined by one or more of the following:

  * serum M-protein concentration ≥ 1 g/dL (10 g/L)
  * urine monoclonal light chain concentration ≥ 200 mg/24 hours as determined by urine protein electrophoresis
  * involved serum free light chain (SFLC) concentration ≥ 10 mg/dL (100 mg/L) and an abnormal SFLC ratio
* Have adequate organ function including:

  * Absolute neutrophil count (ANC) ≥ 1000/microliter
  * Platelet (PLT) count ≥ 75,000/microliter
  * Hemoglobin (Hgb) ≥ 8.0 g/dL
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (if total is elevated check direct and, if normal, participant is eligible)
  * Aspartate transaminase (AST) and alanine aminotransferase (ALT) are ≤ 3 x ULN
  * Serum creatinine ≤ 3.0 mg/dL.
* Have an Eastern Cooperative Oncology Group performance status (ECOG PS) score of ≤ 2.
* Have discontinued all previous therapies for cancer, including chemotherapy, surgery, and radiotherapy for at least 2 weeks (6 weeks for mitomycin-C or nitrosoureas) before study enrollment and recovered from the acute effects of therapy.
* Males and females with reproductive potential: Must agree to use medically approved contraceptive precautions during the study and for 4 months following the last dose of study drug.
* Females with childbearing potential: Must have had a negative urine or serum pregnancy test <7 days before the first dose of study drug.
* Have an estimated life expectancy of ≥16 weeks, in the opinion of the investigator.

Exclusion Criteria:

* Have received treatment within 30 days of the initial dose of study drug with an experimental agent for non-cancer indications that has not received regulatory approval for any indication.
* Have one or more serious preexisting medical conditions that, in the opinion of the investigator, would preclude participation in this study.
* Have an uncontrolled infection.
* Females who are pregnant or breastfeeding.
* Have known positive test results for human immunodeficiency virus (HIV), hepatitis B*, or hepatitis C antibodies (HCAb).

  * Have evidence of or test positive for hepatitis B. A positive test for hepatitis B is defined as:
  1. positive for hepatitis B surface antigen (HBsAg+). OR
  2. positive for anti-hepatitis B core antibody and positive for hepatitis B deoxyribonucleic acid (HBV DNA).

     OR
  3. positive for anti-hepatitis B surface antibody (HBsAb+) and positive for hepatitis B deoxyribonucleic acid (HBV DNA).
* Have ≥ Grade 2 peripheral neuropathy or any grade with pain as assessed using the Common Terminology Criteria for Adverse Events, version 4.03 (CTCAE v 4.03).
* Have previously received an allogenic hematopoietic stem cell transplant.
* Have previously received treatment with an experimental agent that targets B-cell activating factor (BAFF).
* Have a corrected QT (QTc) interval >470 msec on their baseline electrocardiogram (ECG).
* Have interstitial pneumonitis (interstitial pneumonia) or pulmonary fibrosis manifested as opacity on chest X-ray or computed tomography (CT) scan.
* Have had another active malignancy within the past 5 years.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-07; Primary Completion 2015-02 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- Japan (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

REFERENCES:
- [Derived] Iida S, Ogiya D, Abe Y, Taniwaki M, Asou H, Maeda K, Uenaka K, Nagaoka S, Ishiki T, Conti I, Tobinai K. Dose-escalation study of tabalumab with bortezomib and dexamethasone in Japanese patients with multiple myeloma. Cancer Sci. 2016 Sep;107(9):1281-9. doi: 10.1111/cas.13000. Epub 2016 Sep 1. PMID 27350068

RESULTS

PARTICIPANT FLOW:
Groups:
- 100 mg Tabalumab+BTZ IV+Dex: Cohort 1. 100 mg tabalumab (LY2127399)intravenously (IV) on day 1 of each cycle. Bortezomib (BTZ), 1.3 milligram per square meter (mg/m^2), IV on days 1, 4, 8, 11 of Cycle 1-8, then on days 1, 8, 15, 22 from Cycle 9 onward. Oral dexamethasone (Dex), 20 mg/day, on day of and day after BTZ.
- 300 mg Tabalumab+ BTZ +Dex: Cohort 2. 300 mg tabalumab (LY2127399) IV on day 1 of each cycle. BTZ, 1.3 mg/m^2, IV on days 1, 4, 8, 11 of Cycle 1-8, then on days 1, 8, 15, 22 from Cycle 9 onward. Oral dex, 20 mg/day, on day of and day after BTZ subcutaneously or intravenously (SC, IV respectively).
Period: Overall Study
Arm/Group | 100 mg Tabalumab+BTZ IV+Dex | 300 mg Tabalumab+ BTZ +Dex
Started | 4 | 12
Received at Least 1 Dose of Study Drug | 4 (100 mg tabalumab IV) | 12 (300 mg tabalumab IV)
Received BTZ IV | 4 | 4
Received BTZ SC | 0 | 8
Completed | 0 | 1
Not Completed | 4 | 11
Not completed — Adverse Event | 4 | 2
Not completed — Sponsor Decision | 0 | 2
Not completed — Progressive Disease | 0 | 6
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug. 300 mg LY2127399 group administered BTZ IV or SC data were combined per protocol, BTZ was a supplemental therapy for participants.
Groups:
- 100 mg Tabalumab+BTZ IV+Dex: Cohort 1. 100 mg tabalumab (LY2127399) intravenously (IV) on day 1 of each cycle. Bortezomib (BTZ), 1.3 milligram per square meter (mg/m^2), IV on days 1, 4, 8, 11 of Cycle 1-8, then on days 1, 8, 15, 22 from Cycle 9 onward. Oral dexamethasone (Dex), 20 mg/day, on day of and day after BTZ.
- 300 mg Tabalumab+BTZ +Dex: Cohort 2. 300 mg tabalumab (LY2127399) IV on day 1 of each cycle. BTZ, 1.3 mg/m^2, IV on days 1, 4, 8, 11 of Cycle 1-8, then on days 1, 8, 15, 22 from Cycle 9 onward. Oral dex, 20 mg/day, on day of and day after BTZ subcutaneously or intravenously (SC, IV respectively).
- Total: Total of all reporting groups
Arm/Group | 100 mg Tabalumab+BTZ IV+Dex | 300 mg Tabalumab+BTZ +Dex | Total
Number analyzed (Participants) | 4 | 12 | 16
Age, Continuous [Mean (Full Range); unit: years] | 70.7 [66.4 to 80.2] | 71.3 [52.0 to 82.1] | 71.1 [52.0 to 82.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 10
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 12 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 12 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 4 | 12 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Drug Related Adverse Events (AEs) or Any Serious AEs
Description: A summary of other non-serious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline through 8 months
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 100 mg Tabalumab+BTZ IV+Dex | 300 mg Tabalumab+BTZ +Dex
Number analyzed (Participants) | 4 | 12
Participants | 4 | 12

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Plasma Concentration (Cmax) for Tabalumab (LY2127399)
Time Frame: Cycle 1, Day 1: 6 + or - hours after bortezomib (BTZ); Cycle 7, Day 1: immediately post BTZ dose and 2 hours after tabalumab
Population: All participants who received at least 1 dose of any study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (μg/mL)
Groups:
- 300 mg Tabalumab+ IV BTZ +Dex: Cohort 2. 300 mg tabalumab (LY2127399) IV on day 1 of each cycle. BTZ, 1.3 mg/m^2, IV on days 1, 4, 8, 11 of Cycle 1-8, then on days 1, 8, 15, 22 from Cycle 9 onward. Oral dex, 20 mg/day, on day of and day after BTZ IV.
- 300 mg Tabalumab+ SC BTZ +Dex: Cohort 2. 300 mg tabalumab (LY2127399) IV on day 1 of each cycle. BTZ, 1.3 mg/m^2, IV on days 1, 4, 8, 11 of Cycle 1-8, then on days 1, 8, 15, 22 from Cycle 9 onward. Oral dex, 20 mg/day, on day of and day after BTZ SC.
Arm/Group | 100 mg Tabalumab+BTZ IV+Dex | 300 mg Tabalumab+ IV BTZ +Dex | 300 mg Tabalumab+ SC BTZ +Dex
Number analyzed (Participants) | 4 | 4 | 8
microgram per milliliter (μg/mL)
  Cycle 1 Day 1 | 38.5 (12) | 154 (21) | 139 (14)
  Cycle 7 Day 1: number analyzed (Participants) | 1 | 1 | 3
  Cycle 7 Day 1 | 70.5 (NA) — N of 1, Individual data presented, no CV value. | 179 (NA) — N of 1, Individual data presented, no CV value. | 220 (25)

3. Secondary Outcome: Pharmacokinetics (PK): Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measurable Plasma Concentration (AUC0-tlast) of Tabalumab (LY2127399)
Time Frame: as for outcome 2
Population: All participants who received at least 1 dose of any study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours times nanograms per milliliter
Groups:
- 100 mg Tabalumab+BTZ IV+Dex: Cohort 1. 100 mg tabalumab (LY2127399) intravenously (IV) on day 1 of each cycle. Bortezomib (BTZ), 1.3 milligram per square meter (mg/m^2), IV on days 1, 4, 8, 11 of Cycle 1-8, then on days 1, 8, 15, 22 from Cycle 9 onward. Oral dexamethasone (Dex), 20 mg/day, on day of and day after BTZ.
  LY2127399: Administered IV
  Bortezomib IV: Administered IV
  Dexamethasone: Administered orally
- 300 mg Tabalumab IV BTZ +Dex: Cohort 2. 300 mg tabalumab (LY2127399) IV on day 1 of each cycle. BTZ, 1.3 mg/m^2, IV on days 1, 4, 8, 11 of Cycle 1-8, then on days 1, 8, 15, 22 from Cycle 9 onward. Oral dex, 20 mg/day, on day of and day after BTZ IV.
Arm/Group | 100 mg Tabalumab+BTZ IV+Dex | 300 mg Tabalumab IV BTZ +Dex | 300 mg Tabalumab+ SC BTZ +Dex
Number analyzed (Participants) | 4 | 4 | 8
hours times nanograms per milliliter
  Cycle 1 Day 1 | 8100 (15) | 34600 (23) | 26900 (48)
  Cycle 7 Day 1: number analyzed (Participants) | 1 | 1 | 3
  Cycle 7 Day 1 | 9400 (NA) — N of 1, Individual data presented, no CV value. | 27300 (NA) — N of 1, Individual data presented, no CV value. | 22900 (71)

4. Secondary Outcome: Pharmacokinetics (PK): Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-∞) of Tabalumab (LY2127399)
Time Frame: as for outcome 2
Population: All participants who received at least 1 dose of any study drug and had evaluable PK data. Participants in the 300 mg tabalumab group may have received IV and SC BTZ and may be counted in the IV and SC group for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | 100 mg Tabalumab+BTZ IV+Dex | 300 mg Tabalumab+ IV BTZ +Dex | 300 mg Tabalumab+ SC BTZ +Dex
Number analyzed (Participants) | 4 | 4 | 8
ng*hr/mL
  Cycle 1 Day 1 | 13300 (21) | 64200 (35) | 50900 (60)
  Cycle 7 Day 1: number analyzed (Participants) | 1 | 1 | 3
  Cycle 7 Day 1 | NA (NA) — N of 1, no value obtained, no CV value. | 84100 (NA) — N of 1, Individual data presented, no CV value. | 131000 (NA) — CV not available from N=3 for analysis.

5. Secondary Outcome: Number of Participants With Tumor Response (Tumor Response Rate)
Description: Stringent Complete Response- Complete response in addition to normal free light chain ration and no clonal cells in bone marrow.
  Complete Response- no monoclonal protein (mp) in blood, no serum or urine mp, less than 5% plasma cells in bone marrow.
  Very Good Partial Response-more than 90% decrease in mp and urine protein. Partial Response- over 50% decrease in serum mp. Stable Disease- less than 25 percent decrease of monoclonal protein. Progressive Disease- 25% increase compared to lowest value of serum mp, urine mp, no measurable mp.
Time Frame: Baseline to disease progression (up to 421 days)
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- 300 mg Tabalumab+ IV BTZ +Dex: Cohort 2. 300 mg tabalumab (LY2127399) IV on day 1 of each cycle. BTZ, 1.3 mg/m^2, IV on days 1, 4, 8, 11 of Cycle 1-8, then on days 1, 8, 15, 22 from Cycle 9 onward. Oral dex, 20 mg/day, on day of and day after BTZ subcutaneously or intravenously (SC, IV respectively).
Arm/Group | 100 mg Tabalumab+BTZ IV+Dex | 300 mg Tabalumab+ IV BTZ +Dex
Number analyzed (Participants) | 4 | 12
Participants
  Numbers of Responders | 4 | 5
  Stringent Complete Response (sCR) | 0 | 0
  Complete Response (CR) | 0 | 0
  Very Good Partial Response (VGPR) | 2 | 1
  Partial Response(PR) | 2 | 4
  Stable Disease(SD) | 0 | 2
  Progressive Disease | 0 | 3

6. Secondary Outcome: Duration of Response (DoR)
Description: DoR is defined as the time from the date when the measurement criteria are met for CR, CRu, or PR (whichever status is recorded first) until the date of first observation of measured progressive disease. For responding participants who die without progressive disease (including death from study disease),DoR will be censored at the date of death. For responding participants not known to have died as of the data cut-off date and who do not have progressive disease, DoR will be censored at the last objective progression-free assessment date prior to the data cut-off date.
Time Frame: Time from Response until measured Progressive Disease (up to 455 days)
Population: All participants who received at least 1 dose of study drug, 4 participants were censored from Cohort 1 and 5 participants from Cohort 2. 300 mg tabalumab group administered BTZ IV or SC data were combined per protocol, BTZ was a supplemental therapy for participants.
Measure: Number; unit: months
Groups:
- 300 mg Tabalumab+BTZ +Dex: Cohort 2. 300 mg tabalumab (LY2127399) IV on day 1 of each cycle. BTZ, 1.3 mg/m^2, IV on days 1, 4, 8, 11 of Cycle 1-8, then on days 1, 8, 15, 22 from Cycle 9 onward. Oral dex, 20 mg/day, on day of and day after BTZ IV or SC.
Arm/Group | 100 mg Tabalumab+BTZ IV+Dex | 300 mg Tabalumab+BTZ +Dex
Number analyzed (Participants) | 4 | 5
months | NA — Data is not available to be presented because endpoint was not reached. | NA — Data is not available to be presented because endpoint was not reached.

7. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the time from the date of study enrollment to the date of objectively determined progressive disease. TTP will be censored at the date of the last objective progression free disease assessment.
Time Frame: Baseline to date of Progressive Disease (up to 455 days)
Population: All participants who received at least 1 dose of study drug and didn't have AEs . 300 mg tabalumab group administered BTZ IV or SC data were combined per protocol, BTZ was a supplemental therapy for participants. Participants that were censored prior to PD and not included in analysis:100 mg tabalumab n=4, 300 mg tabalumab n=8.
Measure: Median (Full Range); unit: months
Arm/Group | 100 mg Tabalumab+BTZ IV+Dex | 300 mg Tabalumab+BTZ +Dex
Number analyzed (Participants) | 4 | 12
months | NA [NA to NA] — No data collected due to censoring prior to PD. | NA [0.49 to 8] — Due to censoring prior to PD, median not collected as per Statistical Analysis Plan.

8. Secondary Outcome: Pharmacodynamics (PD): Change From Baseline in Absolute B-cell Count
Time Frame: Baseline through study completion (up to 455 days)
Population: Zero participants analyzed as no post baseline data collected.
Groups:
- 100 mg Tabalumab+BTZ IV+Dex: Cohort 1. 100 mg tabalumab (LY2127399)intravenously (IV) on day 1 of each cycle. Bortezomib (BTZ), 1.3 milligram per square meter (mg/m^2), IV on days 1, 4, 8, 11 of Cycle 1-8, then on days 1, 8, 15, 22 from Cycle 9 onward. Oral dexamethasone (Dex), 20 mg/day, on day of and day after BTZ.
  Bortezomib IV: Administered IV
  Dexamethasone: Administered orally
Arm/Group | 100 mg Tabalumab+BTZ IV+Dex | 300 mg Tabalumab+BTZ +Dex
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Pharmacodynamics (PD): Change From Baseline in B-cell Subset Fractions
Description: CD19+ peripheral B-cells counts are based on the percentage of total leukocyte population and absolute cell counts.
Time Frame: Baseline, Cycle 1 and Cycle 7: prior to first tabalumab dose.
Population: All participants who received at least 1 dose of study drug and had evaluable PD. 300 mg tabalumab IV and SC dose were analyzed together.
Measure: Mean (Standard Deviation); unit: percentage of b-cell change
Groups:
- 300 mg Tabalumab+BTZ IV+Dex: Cohort 2. 300 mg tabalumab (LY2127399) IV on day 1 of each cycle. BTZ, 1.3 mg/m^2, IV on days 1, 4, 8, 11 of Cycle 1-8, then on days 1, 8, 15, 22 from Cycle 9 onward. Oral dex, 20 mg/day, on day of and day after BTZ subcutaneously or intravenously (SC, IV respectively).
Arm/Group | 100 mg Tabalumab+BTZ IV+Dex | 300 mg Tabalumab+BTZ IV+Dex
Number analyzed (Participants) | 4 | 12
percentage of b-cell change
  Baseline | 9.3 (8.1) | 12.5 (10.7)
  Cycle 1, Day 1 | 1.1 (1.6) | 0.3 (6.7)
  Cycle 7, Day 1: number analyzed (Participants) | 1 | 4
  Cycle 7, Day 1 | NA (NA) — N of 1, pd data not collected from participant | -14.4 (7.5)

ADVERSE EVENTS:
Description: 300 mg tabalumab (LY2127399) group administered BTZ IV or SC data were combined per protocol, BTZ was a supplemental therapy for participants.
Arm/Group | 100 mg Tabalumab+BTZ IV+Dex | 300 mg Tabalumab+BTZ +Dex
Serious Adverse Events (participants affected / at risk) | 2/4 | 8/12
Other Adverse Events (participants affected / at risk) | 4/4 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 mg Tabalumab+BTZ IV+Dex (N=4) | 300 mg Tabalumab+BTZ +Dex (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 mg Tabalumab+BTZ IV+Dex (N=4) | 300 mg Tabalumab+BTZ +Dex (N=12)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 5 (7)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (5) | 5 (8)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (3)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 4 (5)
Injection site erythema (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 2 (3)
Oedema (General disorders) | 0 (0) | 3 (3)
Oedema peripheral (General disorders) | 1 (1) | 2 (2)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (3)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (2) | 2 (3)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 3 (5)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 2 (2)
Blood phosphorus decreased (Investigations) | 1 (2) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 5 (11)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 2 (3) | 4 (9)
Weight decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 3 (6)
White blood cell count increased (Investigations) | 0 (0) | 1 (9)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 4 (6)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (4) | 4 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Dysgeusia (Nervous system disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 3 (3)
Vagus nerve disorder (Nervous system disorders) | 1 (2) | 3 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
300 mg tabalumab (LY2127399) group administered BTZ IV or SC data were combined per protocol in some instances as BTZ was a supplemental therapy for participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days